CLINICAL TRIAL: NCT05371366
Title: A Multicenter, Randomized, Parallel-controlled Clinical Trial to Evaluate the Efficacy and Safety of a New Atrial Septal Defect Occluder, ReAces®, and Delivery System for the Treatment of Atrial Septal Defect Occlusion
Brief Title: The Puncturable Atrial Septal Defect Occluder Trial (the PASSER Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Principal Investigator, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYYL2022-06ZC-01
Record Dates: First submitted 2022-05-04; First posted 2022-05-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients with ASD assigned to experimental group will receive the novel ASD occluder (ReAces)
  Interventions: Device: ASD closure with the novel occluder (ReAces)
- Control Group (Active Comparator): Patients with ASD assigned to control group will receive the normal occluder
  Interventions: Device: ASD closure with normal occluder

INTERVENTIONS:
Device: ASD closure with the novel occluder (ReAces) — Transcatheter closure atrial septal defect with the novel occluder (ReAces)
  Arms: Experimental group
Device: ASD closure with normal occluder — Transcatheter closure atrial septal defect with normal occluder
  Arms: Control Group

SUMMARY:
A multicenter, randomized, parallel-controlled clinical trial to evaluate the efficacy and safety of a new atrial septal defect occluder, ReAces®, and delivery system for the treatment of atrial septal defect occlusion. Compared with the traditional atrial septal occluder, this new atrial septal occluder supports re-puncture after occluder implantation. Thus those patients who have undergone atrial septal defect closure with the novel device may be eligible for future radiofrequency ablation of atrial fibrillation or mitral valve intervention.

The trial is expected to enroll 128 patients who will be randomly assigned to the test group or control group in a 1:1 ratio. Patients in test group will received ReAces occluder，and the others the regular occluder.The experiment is scheduled to enroll 128 patients who will be randomly allocated to one of two groups: test or control. Patients in the test group will receive a ReAces occluder, while those in the control group will receive a standard occluder.The safety and efficacy of the two groups at 1 year after surgery will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-70 years;
2. with congenital secundum atrial septal defect;
3. the maximal ASD diameter was ≤38 mm;
4. with atrial-level left-to-right shunt, with Qp/Qs shunt ratio ≥1.5:1, or TTE or clinical manifestations indicated the existence of defect that inducing overfilling of right atrium;
5. the distance from the margin of defect to coronary sinus, atrioventricular (AV) valve, and right superior pulmonary vein (RSPV) was ≥5 mm, according to the echocardiography measurements;
6. volunteered to participate in this study, and signed informed consents.

Exclusion Criteria:

1. ostium primordium ASD and sinus venosus ASD.
2. infective endocarditis and hemorrhagic disorders.
3. active thrombosis.
4. patients with severe pulmonary hypertension (mean pulmonary artery pressure measured by catheter > 30 mmHg) who are not taking targeted drugs
5. patients with a porous atrial septal defect that cannot be completely occluded by a single occluder.
6. with severe myocardial disorders or valvular disease not associated with ASD
7. infectious disease within the last 1 month, or uncontrolled infectious disease
8. bleeding disorders, untreated gastric or duodenal ulcers
9. thrombosis in left atrium
10. partial or total pulmonary vein ectopic drainage
11. left atrial septum, left atrial or left ventricular dysplasia
12. Patients whose size (too small for TEE probe, catheter size, etc.) or physical condition (active infection, etc.) makes them unsuitable for cardiac catheterization
13. Patients who are allergic to nickel
14. Patients with any contraindication to aspirin therapy (except for those able to take other antiplatelet agents for 6 consecutive months).
15. Pregnant or lactating women and those who plan to become pregnant during the trial
16. Patients with a life expectancy of <12 months or those who are unable to complete the study's prescribed follow-up schedule
17. Participation in another clinical trial of a drug or medical device within 30 days prior to screening.
18. Patients who have previously undergone surgical atrial septal defect repair or percutaneous interventional atrial septal defect closure.
19. Patients who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-04-22 (Estimated); Study Completion 2023-04-22 (Estimated)

PRIMARY OUTCOMES:
Successful rate of complete closure of atrial septal defect | 0-360 days
  The success rate of complete closure at 12 months after the procedure was used as the main efficacy index to evaluate the effectiveness of the novel atrial septal defect occluder ReAces, reflecting the long-term implantation effect of the device.

SECONDARY OUTCOMES:
Adverse events | 0-360 days
  all cause and cardiovascular mortality, pericardial tamponade, cerebrovascular events, malignant arrhythmia, infection, device migration, and occluder-related thrombosis or embolization during the operation or follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fang Y, Hou K, Lin D, Zhou D, Pan W, Ge J. Device endothelialization and morphology assessments at 1 year using computed tomography angiography: comparison of traditional with novel puncturable atrial septal defect occluders. BMC Cardiovasc Disord. 2024 Dec 30;24(1):755. doi: 10.1186/s12872-024-04438-1. PMID 39734195